CLINICAL TRIAL: NCT03688451
Title: A Pilot Study to Access the Feasibility and Safety of Intrathecal Rituximab Added to Standard Intrathecal Prophylaxis to Prevent CNS Relapse for CD 20 Positive Non Hodgkin Lymphoma
Brief Title: Intrathecal Rituximab With Standard Intrathecal Prophylaxis to Prevent CNS Relapse for CD 20+ Non Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tahir Latif (Other)
Responsible Party: Sponsor-Investigator, Tahir Latif, Professor of Medicine, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UCCI-HEM-17-01
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: Sequential dose cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intrathecal rituximab (Experimental): Cohort 1: 10 mg dose, day 1 chemotherapy cycles 2-5 Cohort 2: 20 mg dose, day 1 chemotherapy cycles 2-5
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Intrathecal administration over 3-5 minutes

SUMMARY:
The purpose of this research study is to learn if giving rituximab, the study drug, right into the spinal canal along with chemotherapy drugs like methotrexate is possible and safe.

ELIGIBILITY:
Inclusion Criteria:

* CD20 positive diffuse large b-cell lymphoma undergoing treatment with systemic rituximab in combination with CHOP, CHOEP, or EPOCH and deemed high risk of CNS relapse and eligible for central nervous system prophylaxis with intrathecal therapy.

Exclusion Criteria:

* Primary central nervous system lymphoma or established secondary central nervous system disease.
* History of spinal surgery and/or ineligible for intrathecal injections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-29 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Ability to deliver greater than 80% of planned doses | 28 months
  Percentage of planned doses administered for planned accrual
Related Grade 3 or higher non-hematological toxicity | 28 months
  Number of related grade 3 or higher non-hematological toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Tahir Latif, MD, Principal Investigator — University of Cincinnati
Locations (1):
- UC Health, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No